CLINICAL TRIAL: NCT06710912
Title: The Effectiveness of Group Acceptance and Commitment Therapy (ACT) Among Mild to Moderate Depressive Patients in Kelantan, Malaysia
Brief Title: Group Acceptance and Commitment Therapy (ACT) Among Depressive Patients in Kelantan, Malaysia
Acronym: Group ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Aisyah Che Rahimi, Dr, Universiti Sains Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USM/JEPeM/22040192; 304/PPSP/6315752 (Other Grant/Funding Number: Universiti Sains Malaysia)
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: acceptance and commitment therapy (ACT); group therapy; depression; psychological flexibility; quality of life
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants in the ACT group attended four sessions of Acceptance and Commitment Therapy over a four-week period with each session lasting around 90-120 minutes. The participants were divided into three subgroups, each of which included approximately 6 to 8 participants. Prior to the intervention, participants in the ACT group received a workbook which consists of information about ACT in summary. Participants in the ACT group had accessibility to the same care similar to the TAU group. Four sessions were held for each subgroup respectively which was conducted by at least two therapists trained in ACT. The ACT module was adapted from Hayes and Harris and were conducted in the Malay language. The same workbook with guided exercise and homework were used by all the therapists to assure standardization of the intervention to ensure that each group received similar contents in each session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ACT (Experimental): Participants of this arm underwent 4 weeks of weekly session of acceptance and commitment therapy (ACT).
  Interventions: Behavioral: Group acceptance and commitment therapy (ACT)
- Treatment-as-usual (TAU) group (Active Comparator): The participants in this group received standard treatment for major depressive disorder
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Group acceptance and commitment therapy (ACT) — The ACT intervention module utilized in this study was adapted from Hayes foundational work on ACT and Harris. A summary of the general contents and exercises in each week was in accordance with the 6 core processes of Acceptance and Commitment Therapy based on Hayes. It was conducted in the Malay language. The same workbook with guided exercise and homework were used by all the therapists to assure standardization of the intervention to ensure that each group received similar contents in each session.
  Arms: Group ACT
Other: Treatment as usual — Standard care and follow-up for major depressive disorder
  Arms: Treatment-as-usual (TAU) group

SUMMARY:
The goal of this clinical trial is to learn if group acceptance and commitment therapy works to improve depressive symptoms, psychological flexibility and quality of life in adults. The main questions it aims to answer are:

1. What is the effectiveness of group Acceptance and Commitment Therapy (ACT) in reducing depressive symptoms among depressive patients in Kelantan from pre- to post-intervention and at 3 months follow-up?
2. What is the mean difference of quality of life among depressive patients in Kelantan who undergo group ACT from pre- to post-intervention and at 3 months follow-up?
3. What is the effectiveness of group ACT in improving the psychological flexibility among depressive patients in Kelantan from pre- to post intervention and at 3 months follow-up?

Researchers will compare group ACT group to a treatment-as-usual (TAU) group to see if group ACT works to improve depressive symptoms, quality of life and psychological flexibility.

Participants will:

* Attend weekly ACT sessions for four weeks or undergo standard treatment for major depressive disorder.
* Fill up four questionnaires before the intervention, after a month and at 3-month follow-up.

DETAILED DESCRIPTION:
General Objectives To study the effectiveness of group Acceptance and Commitment Therapy in the treatment of depression among depressive patients in Kelantan.

Specific Objectives

1. To evaluate the effectiveness of group Acceptance and Commitment Therapy (ACT) in reducing the symptoms of depression in patients in Kelantan from pre- to post-intervention and at 3 months follow-up.
2. To determine the effectiveness of group Acceptance and Commitment Therapy (ACT) in improving the quality of life of patients with depression in Kelantan from pre- to post-intervention and at 3 months follow-up.
3. To assess the effectiveness of group Acceptance and Commitment Therapy (ACT) in improving the psychological flexibility of patients with depression in Kelantan from pre- to post intervention and at 3 months follow-up.

This quasi-experimental study used a two-group design, comparing group ACT with TAU at baseline, post-intervention, and a 3-month follow-up. Conducted at the Psychiatry Clinic, Hospital Universiti Sains Malaysia, from June 2022 to May 2024, the study included 44 participants with mild to moderate depression. Twenty-two participants allocated in the ACT group received weekly group ACT sessions over four weeks, while twenty-two participants were assigned to the TAU group. Outcomes were measured using the Malay versions of the Beck Depression Inventory I (BDI), WHO Quality of Life-BREF (WHOQOL-BREF), and Acceptance and Action Questionnaire II (AAQ-II) at baseline, post-intervention, and at 3-month follow-up. Data was analyzed using two-way Repeated Measures Analysis of Variance (RM ANOVA) to assess changes in these outcomes across the different time points.

ELIGIBILITY:
Inclusion Criteria:

* had a Beck Depression Inventory (BDI) score ranging from 10 to 29, indicating mild to moderate depression.
* Proficient in the Malay language
* Willing to commit to the study.

Exclusion Criteria:

* Have concomitant psychotic symptoms.
* Participated and enrolled in Cognitive Behavioural Therapy.
* previously had participated in Acceptance Commitment Therapy.
* had underlying substance use disorder or active substance use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | From enrollment to the end of treatment at 4 weeks
  The outcome was measured by using Beck Depression Inventory (BDI)
Quality of life | From enrollment to the end of treatment at 4 weeks
  The outcome was measured by using brief WHO Quality of Life (WHOQOL) questionnaire (Malay version)
Psychological flexibility | From enrollment to the end of treatment at 4 weeks
  The outcome was measured using Acceptance and Action Questionnaire II Malay Version (AAQ-II)

SECONDARY OUTCOMES:
Depressive symptoms (3 months) | 3 months post intervention
  It was measured using BDI at 3 months post-intervention
Quality of life (3 months) | 3 months post intervention
  It was measured using WHOQOL at 3 months post-intervention
Psychological flexibility (3 months) | 3 months post intervention
  It was measured using AAQ-II at 3 months post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rong J, Cheng P, Li D, Wang X, Zhao D. Global, regional, and national temporal trends in prevalence for depressive disorders in older adults, 1990-2019: An age-period-cohort analysis based on the global burden of disease study 2019. Ageing Res Rev. 2024 Sep;100:102443. doi: 10.1016/j.arr.2024.102443. Epub 2024 Aug 7. PMID 39097004